CLINICAL TRIAL: NCT06913218
Title: An Exploratory Study to Evaluate Safety and Efficacy of the Neoantigen Personalized mRNA Vaccine AK154 Monotherapy or in Combination With AK104 or AK112,and the Sequential mFOLFIRINOX Regimen as Adjuvant Therapy in Surgically Resectable Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of mRNA Vaccines AK154 Monotherapy or in Combination With AK104/AK112,and Sequential mFOLFIRINOX in Surgically Resected PDAC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK154-IIT-001
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Cancer; Pancreas Cancer, Duct Cell Adenocarcinoma
Keywords: adjuvant; pancreas cancer; mRNA
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pancreatic Cancer (Experimental): Resectable PDAC
  Interventions: Biological: AK154; Biological: Cadonilimab; Biological: Ivonescimab (SMT112 or AK112) Injection; Drug: mFOLFORINOX

INTERVENTIONS:
Biological: AK154 — AK154 is neotigeon personalized mRNA vaccine
Biological: Cadonilimab — a PD-1/CTLA-4 bispecific antibody
Biological: Ivonescimab (SMT112 or AK112) Injection — a PD-1/VEGF bi-specific antibody
Drug: mFOLFORINOX — mFOLFIRINOX:Fluorouracil+leucovorin+Irinotecan+Oxaliplatin

SUMMARY:
To explore safety and efficacy of neoantigen personalized mRNA vaccines AK154 monotherapy or in combination with AK104/AK112 and sequential mFOLFIRINOX regime in Resected PDAC

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center, exploratory clinical study. To explore the safety, tolerability, efficacy, immunogenicity, and PK/PD profile of neoantigen personalized mRNA vaccine AK154 monotherapy or combined with AK104 or AK112, sequential mFOLFIRINOX chemotherapy regimen as postoperative adjuvant therapy in Surgically Resected Pancreatic Adenocarcino

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed the informed consent form and complied with protocols requirements
* Patients with radiographically resectable primary pancreatic tumors
* Histopathology or cytology confirmed resected PDAC with macroscopic complete resection (R0 and R1)
* Pancreatic cancer surgical staging per AJCC 8th edition staging: T 1-3, N0-2, M0
* ECOG 0 or 1
* Life expectancy ≥ 6 months
* Surgical complications have recovered,
* Adequate organ function
* Patients with fertility are willing to use an adequate method of contraception.

Exclusion Criteria:

* The presence of other pathologic types
* Participating in another clinical study
* Have received treatment for pancreatic cancer, including chemotherapy, radiation therapy, targeted therapy, immunotherapy,etc
* Plan to receive a live-attenuated vaccine within 28 days prior to initiation of study treatment or during the study treatment or within 90 days after the end of study treatment
* Severe infection occurs within 4 weeks prior to the first dose
* Requiring systemic therapy with glucocorticoids or other immunosuppressive drugs within 14 days prior to initial administration.
* Acute pancreatitis or subclinical pancreatitis
* Active autoimmune disease
* Allergic to immunotherapies and related drugs
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Splenectomy history
* Active tuberculosis
* Known or highly suspected history of interstitial pneumonia.
* Clinically significant liver disease
* Uncontrolled or severe cardiovascular disease.
* Severe bleeding tendency or history of coagulopathy
* Active malignancy within the last 3 years
* Active syphilis infection
* Any other situations that are not suitable for inclusion in this study judged by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2028-02-23 (Estimated); Study Completion 2028-11-06 (Estimated)

PRIMARY OUTCOMES:
DLT | Day 1 to Day 21 after the first tumour vaccine was administrated
  Percentage of subjects who meet the criteria of DLT in DLT observation period
AE | From ICF up to 30days after last study treatment
  Percentage of subjects with Adverse Events (AEs)

SECONDARY OUTCOMES:
RFS | 2 years
  Recurrence free survival（RFS）
OS | 2 years
  Overall survival（OS）

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery,Fudan University Shanghai Cancer Center, Shanghai, Xuhui, China

IPD SHARING:
Plan to Share IPD: Undecided